CLINICAL TRIAL: NCT04946370
Title: Phase I/II Trial of Pembrolizumab and Androgen-receptor Inhibitor With or Without 225Ac-J591 for Progressive Metastatic Castration Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-08022500
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pembrolizumab; Androgen Receptor Antagonists

STUDY DESIGN:
Intervention Model Description: In the phase I portion of the study, patients will receive 225Ac-J591 at either 65 or 80 KBq/kg, in addition to pembrolizumab and ARI. In the subsequent phase II portion of the study, patients will be randomized to receive 225Ac-J591 (at the dose determined in phase I) + ARI and pembrolizumab or ARI and pembrolizumab alone in a 1:1 ratio. Randomization will take into account prior receipt of ARI, baseline PSMA imaging intensity, and presence of visceral metastasis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + 225Ac-J591 + ARI (Experimental): Patients will receive one dose of 225Ac-J591 (single dose, either 65 or 80 Kbq/kg) in combination with pembrolizumab (400mg every 6 weeks) and ARI (standard dose schedule, examples of ARI include enzalutamide, apalutamide, darolutamide).
  Interventions: Drug: 225Ac-J591; Drug: Pembrolizumab; Drug: Androgen receptor inhibitor; Diagnostic Test: 68Ga-PSMA-11
- Pembrolizumab + ARI (Experimental): Patients will receive pembrolizumab (400mg every 6 weeks) and ARI (standard dose schedule) without 225Ac-J591.
  Interventions: Drug: Pembrolizumab; Drug: Androgen receptor inhibitor; Diagnostic Test: 68Ga-PSMA-11

INTERVENTIONS:
Drug: 225Ac-J591 — Alpha-emitter Actinium-225 conjugated to the anti-PSMA antibody J591.
  Arms: Pembrolizumab + 225Ac-J591 + ARI
Drug: Pembrolizumab — Pembrolizumab will be administered intravenously, 400mg every 6 weeks. Patients may receive maximum 18 cycles of therapy, approximately 2 years.
Drug: Androgen receptor inhibitor — Patients will receive an oral androgen receptor inhibitor (ARI). Examples include enzalutamide, apalutamide, darolutamide. Dosing will be the standard dosing, as described by the package insert.
Diagnostic Test: 68Ga-PSMA-11 — [185 ±74 MBq or 5 ±2 mCi] intravenous during screening and 12 weeks. Imaging agent for PSMA PET/CT.
  Other Names: 68Ga-PSMA-HBED-CC

SUMMARY:
This is a phase I/II study investigating the combination of 225Ac-J591 (a drug that can deliver radiation to prostate cancer cells) with pembrolizumab (immunotherapy, a drug that increases the immune system's ability to destroy cancer cells). This study will assess whether 225Ac-J591 + pembrolizumab + androgen receptor inhibitor (ARI) is more effective against prostate cancer than pembrolizumab + ARI alone.

DETAILED DESCRIPTION:
This clinical trial is for men with progressive metastatic castration-resistant prostate cancer (mCRPC). The primary objectives of the study are to determine the optimal dose of 225Ac-J591 when combined with pembrolizumab (phase I) and then to assess whether the combination of 225Ac-J591, pembrolizumab, and androgen receptor inhibitor (ARI) is more effective against prostate cancer than pembrolizumab and ARI alone. 225Ac-J591 is a radionuclide conjugate involving Actinium-225 linked to J591, an antibody that recognizes prostate-specific membrane antigen (PSMA) on the surface of cancer cells; 225Ac-J591 is able to deliver powerful radiation to cancer cells. Pembrolizumab is a drug that strengthens the body's immune response to cancer cells.

In the phase I portion of the study, two cohorts of up to 6 patients each will receive combined therapy: ARI (standard dosing schedule), pembrolizumab (400 mg every 6 weeks), 225Ac-J591 (single dose, either 65 or 80 KBq/kg). Following a minimum of 12 weeks of safety follow-up, the study team will determine which 225Ac-J591 dose is better.

In the phase II portion, patients will be randomized to pembrolizumab + ARI with or without 225Ac-J591. The primary endpoint for phase II will be response - a composite of PSA, circulating tumor cell (CTC) count and imaging changes, comparing baseline and Week 12 measurements. Patients who achieve at least one of the criteria will be considered responders. Imaging (CT scan, bone scan) will occur every 12 weeks. Additionally, participants will undergo 68Ga-PSMA-11 PET/CT scan prior to therapy and at 12 weeks. Patients are able to receive pembrolizumab every 6 weeks for maximum 18 cycles (approximately 2 years).

ELIGIBILITY:
Inclusion Criteria:

* Male participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of prostate adenocarcinoma.
* A male participant must agree to use a contraception during the treatment period and for at least 4 months after the last dose of study treatment and refrain from donating sperm during this period.
* Documented progressive metastatic CRPC based on Prostate Cancer Working Group 3 (PCWG3) criteria, which includes at least one of the following criteria: PSA progression, Objective radiographic progression in soft tissue, New bone lesions
* Evaluable for response with at least one of the following:

  * Measurable disease by RECIST 1.1
  * Detectable (>0) CTC by CellSearch
  * PSA of at least 5ng/dL
* ECOG performance status of 0-1
* Have serum testosterone ≤ 50 ng/dL. Subjects must continue primary androgen deprivation with an LHRH/GnRH analogue (agonist/antagonist) if they have not undergone orchiectomy.
* Have previously been treated with at least one of the following in any disease state: Androgen receptor inhibitor (ARI, such as enzalutamide, apalutamide or darolutamide), CYP 17 inhibitor (such as abiraterone acetate). These drugs may have been initiated in the metastatic hormone sensitive (i.e. non-castrate) or non-metastatic (M0) CRPC setting provided they meet criteria for progressive mCRPC at study entry.
* Age ≥ 18 years
* Patients must have normal organ and marrow function as defined: Absolute neutrophil count >2,000 cells/mm3, Hemoglobin ≥ 9 g/dL, Platelet count >150 x 10^3/mcL, Serum creatinine <1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 50 mL/min/1.73 m2 by Cockcroft-Gault, Serum total bilirubin <1.5 x ULN (unless due to Gilbert's syndrome in which case direct bilirubin must be normal), Serum AST and ALT <3 x ULN in absence of liver metastases; < 5x ULN if due to liver metastases (in both circumstances bilirubin must meet entry criteria), Serum internalized normalized ratio (INR) OR prothrombin time (PT) AND activated partial thromboplastin time (aPTT) must be ≤1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior receipt of chemotherapy for castration-resistant prostate cancer. Prior receipt of docetaxel chemotherapy in the hormone sensitive setting or for localized disease is acceptable provided at least 6 months has passed since the last dose.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* Prior bone-seeking beta-emitting radioisotopes (e.g. Sm-153, Sr-89) or PSMA-targeted radionuclide therapy for metastatic disease; prior radium-223 is allowed provided last dose administered >12 weeks prior to C1D1 on this study
* Has a history of a second malignancy, unless treatment with curative intent has been completed with no evidence of malignancy for 2 years. Patients with treated localized non-melanoma skin care, non-muscle invasive urothelial carcinoma, or carcinoma in-situ of other site are not excluded.
* Known history of myelodysplastic syndrome
* Has a known history of Human Immunodeficiency Virus (HIV) infection
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks or <5 half-lives prior to enrollment.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
* Diagnosis of deep vein thrombosis and/or pulmonary embolus within 1 month of C1D1
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has received radiotherapy within 4 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation to non-CNS disease that is not a measurable target lesion.
* Patients on stable dose of bisphosphonates or denosumab, which have been started no less than 4 weeks prior to treatment start, may continue on this medication, however patients are not allowed to initiate bisphosphonate/denosumab therapy during the DLT-assessment period of the study. These drugs may be added after week 12 in phase 1 or phase 2.
* Unless azoospermia is present (whether due to surgery or underlying medical condition), having partners of childbearing potential and not willing to use a method of birth control deemed acceptable by the principal investigator and chairperson during the study and for 4 months after last study drug administration.
* Is expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines are allowed.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy at the time of treatment initiation
* Has a known history of active TB (Bacillus Tuberculosis)
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Has had an allogenic tissue/solid organ transplant

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Metastatic Castrate Resistant Prostate Cancer
Enrollment: 37 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with dose-limiting toxicity (DLT) following treatment with pembrolizumab and 225Ac-J591 | From visit 1 through 12 weeks on study
  Primary outcome for phase I; DLTs will be measured by utilizing the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. There will be 12 weeks of safety follow-up following visit 1.
Determination of optimal dose of 225Ac-J591 for phase II | From visit 1 through 12 weeks on study
  Primary outcome for phase I; following 12 weeks of safety follow-up, the study team will make a determination of the 225Ac-J591 dose for phase II (either 65 or 90 KBq/kg).
Change in composite response rate of pembrolizumab and ARPI with or without 225Ac-J591 | Will be collected at the time of visit 1 and up to 100 months
  The primary outcome for phase II will be response, a composite of: PSA decline greater than 50% of baseline, measurable disease response by imaging criteria, conversion of circulating tumor cell count to favorable or undetectable.

SECONDARY OUTCOMES:
Change in overall survival following treatment | Survival will be collected from Day 1 and up to 100 months
  Overall survival will be captured through in-clinic or telephone contact with subjects
Change in biochemical progression-free survival | Will be collected at the time of visit 1 and up to 100 months
  PSA progression will be defined as a rise of > 25% above either the pretreatment level or the nadir PSA level (whichever is lowest). PSA must increase by > 2 ng/ml to be considered progression.
Change in radiographic progression-free survival | Patients will undergo imaging at screening and then every 12 weeks, for up to 100 months
  Response evaluation criteria in solid tumors RECIST (Version 1.1) criteria with prostate cancer working group 3 (PCWG3) modifications will be used.
Change in proportion with 1-year progression-free survival | Will be collected at the time of visit 1 through 1 year on study
  By imaging (RECIST 1.1 criteria with prostate cancer working group 3 modifications) or biochemical (PSA) criteria
Change in proportion with >30% PSA decline | Will be collected at the time of visit 1 and up to 100 months
  Baseline (pre-treatment) PSA levels will be compared to PSA nadir on study
Change in proportion with >50% PSA decline | Will be collected at the time of visit 1 and up to 100 months
  Baseline (pre-treatment) PSA levels will be compared to PSA nadir on study
Change in proportion with >90% PSA decline | Will be collected at the time of visit 1 and up to 100 months
  Baseline (pre-treatment) PSA levels will be compared to PSA nadir on study

CONTACTS AND LOCATIONS:
Overall Officials: Scott Tagawa, MD, MS, Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - New York Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - New York Presbyterian/Weill Cornell Medical Center, New York, New York
  - Columbia University Irving Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No